CLINICAL TRIAL: NCT05105477
Title: Hypotension Prediction Index (HPI) Software Guided Hemodynamic Management for Noncardiac Surgery Patients - Blood Pressure Trial (National PI: Kamal Maheshwari, MD, MPH)
Brief Title: Hypotension Prediction Index (HPI) SMART-BP Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted prematurely; voluntarily discontinuation of trial as study specific protocol not followed during data collection
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-04
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Moderate to High-risk Noncardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HPI Arm (Experimental): AcumenTM HPI Software Feature to guide hemodynamic management in moderate-to-high-risk noncardiac surgery.
  Interventions: Device: AcumenTM HPI Software Feature
- Non-HPI arm (Placebo Comparator): Non-protocolized standard of care management per clinician and provider judgement
  Interventions: Other: Non-protocolized Standard of Care

INTERVENTIONS:
Device: AcumenTM HPI Software Feature — The AcumenTM HPI Feature Software provides the clinician with physiological insight into a patient's likelihood of trending toward a hypotensive event. The AcumenTM HPI Feature Software suite is enabled by the minimally invasive Acumen IQ sensor.
  Arms: HPI Arm
Other: Non-protocolized Standard of Care — Non-protocolized standard of care to treat subjects
  Arms: Non-HPI arm

SUMMARY:
A multicenter, randomized comparison of intraoperative hemodynamic management with or without a protocolized strategy utilizing Hypotension Prediction Index (HPI) software guidance during moderate-to-high-risk noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age >18 years
3. ASA Physical Status > 2
4. Noncardiac surgery with expected surgery duration > 2 hours (example include: orthopedic, spine, urology, and general surgery)
5. Planned blood pressure monitoring with an arterial line catheter;
6. General anesthesia;

Exclusion Criteria:

1. Participating in another interventional Trial;
2. Contraindication to arterial blood pressure monitoring;
3. Subjects with a physical site area too limited for proper Sensor placement
4. Serum creatine > 175 μmol/L (>2.0 mg/dL) or CKD stage > 3A
5. Scheduled for intracranial surgery with permissive hypotension;
6. Patient who is confirmed to be pregnant and/or nursing mothers;
7. Patients with an intra-aortic balloon pump (IABP) or ventricular assist device(s);
8. Have a condition that precludes routine or tight blood pressure management such as surgeon request for relative hypotension;
9. Emergency surgery;
10. Require beach-chair positioning;
11. Scheduled for cardiac surgeries
12. Have previously participated in the SMART-BP trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - UC Davis Medical Center, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Medical Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UT Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the time of study termination, 407 subjects were enrolled, which included 369 pivotal subjects. Data from the pilot subjects were not analyzed for study outcomes. Only 369 subjects were pivotal subjects that were analyzed for study outcomes. The tables below display the information and results from the 369 pivotal subjects.
Groups:
- HPI Arm: Acumen HPI Software Feature: The Acumen HPI Feature Software provides the clinician with physiological insight into a patient's likelihood of trending toward a hypotensive event. The Acumen HPI Feature Software suite is enabled by the minimally invasive Acumen IQ sensor.
Period: Overall Study
Arm/Group | HPI Arm | Non-HPI Arm
Started | 187 | 182
Completed | 157 | 159
Not Completed | 30 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPI Arm | Non-HPI Arm | Total
Number analyzed (Participants) | 187 | 182 | 369
Age, Continuous [Mean (Full Range); unit: years] | 63 [18 to 91] | 63 [22 to 91] | 63 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 77 | 163
  Male | 101 | 105 | 206
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American or Black | 18 | 11 | 29
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Declined to identify | 9 | 6 | 15
  White | 150 | 158 | 308
  Other | 7 | 5 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 187 | 182 | 369

OUTCOME MEASURES:

1. Primary Outcome: A Composite of 30-day Moderate-to-severe Perfusion Related Postoperative Complications.
Description: A composite of 30-day moderate-to-severe perfusion related postoperative complications.
Time Frame: From post non-cardiac surgery to 30 days.
Measure: Number; unit: participants with post-op complications
Arm/Group | HPI Arm | Non-HPI Arm
Number analyzed (Participants) | 157 | 159
participants with post-op complications | 19 | 19

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | HPI Arm | Non-HPI Arm
All-Cause Mortality (participants affected / at risk) | 3/187 | 1/182
Serious Adverse Events (participants affected / at risk) | 48/187 | 38/182
Other Adverse Events (participants affected / at risk) | 19/187 | 21/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPI Arm (N=187) | Non-HPI Arm (N=182)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus Paralytic (Gastrointestinal disorders) | 3 (3) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-Abdominal Fluid Collection (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Unknown Cause Of Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Unknown Cause Of Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Other (Hepatobiliary disorders) | 2 (2) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 3 (3)
Abscess (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Wound Infection (Infections and infestations) | 2 (2) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 1 (1)
Other (Infections and infestations) | 1 (1) | 0 (0)
Mental Status Changes Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Troponin Increased (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1) | 0 (0)
Other (Nervous system disorders) | 2 (3) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 12 (12)
Other (Renal and urinary disorders) | 3 (3) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Abdominal Cavity Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Other (Surgical and medical procedures) | 2 (2) | 1 (1)
Distributive Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock Hemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Other (Vascular disorders) | 3 (3) | 2 (2)
Other (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPI Arm (N=187) | Non-HPI Arm (N=182)
Troponin Increased (Investigations) | 19 (20) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT05105477/Prot_SAP_000.pdf